CLINICAL TRIAL: NCT02104947
Title: A Phase III Case Series Clinical Study of the Reversal of the Anticoagulant Effects of Dabigatran by Intravenous Administration of 5.0g Idarucizumab (BI 655075) in Patients Treated Wtih Dabigatran Etexilate Who Have Uncontrolled Bleeding or Require Emergency Surgery or Procedures.RE-VERSE AD (A Study of the RE-VERSal Effects of Idarucizumab on Active Dabigatran) Trial
Brief Title: Reversal of Dabigatran Anticoagulant Effect With Idarucizumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1321.3; 2013-004813-41 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — idarucizumab

ARMS (1):
- idarucizumab (Experimental): idarucizumab Only 1 treatment, no placebo or comparator
  Interventions: Drug: idarucizumab

INTERVENTIONS:
Drug: idarucizumab — idarucizumab

SUMMARY:
Evaluate the reversal of the anticoagulant effects of dabigatran by IV administration of 5.0g idarucizumab in patients treated with dabigatran etexilate who have uncontrolled bleeding or require emergency surgery or procedures.

ELIGIBILITY:
Inclusion criteria:

* Group A (Bleeding patients)

  * Overt bleeding judged by the physician to require a reversal agent
  * Currently taking dabigatran etexilate
  * At least 18 years of age
  * Written informed consent
* Group B (Patients who are taking dabigatran who may not be bleeding, but do require an emergency surgery or procedure for a condition other than bleeding

  * Condition requiring emergency surgery or invasive procedure where adequate hemostasis is required. Emergency is defined as within the following 8 hours.
  * Current treatment with dabigatran
  * At least 18 years of age
  * Written Informed consent.

Exclusion criteria:

* Group A (Bleeding Patients)

  * Patients with minor bleeds (epistaxis, hematuria) who can be managed with standard supportive care.
  * Patients with no clinical signs of bleeding
  * Contraindications to study medication including known hypersensitivity to the drug or its excipients.
* Group B (Patients who require emergency surgery or procedure)

  * A surgery or procedure which is elective or where the risk of uncontrolled or unmanageable bleeding is low.
  * Contraindications to study medication including known hypersensitivity to the drug or its excipients (subjects with hereditary fructose intolerance may react to sorbitol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2014-05-06 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (176):
- United States (30):
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Gainesville, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Community Hospital, Munster, Indiana
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Henry Ford Allegiance Health, Jackson, Michigan
  - Mercy Hospital St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - St. Elizabeth Youngstown Hospital, Youngstown, Ohio
  - St. John Health System Inc, Tulsa, Oklahoma
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Health Research and Education Institute, Fort Worth, Texas
  - Memorial Hermann Hospital - Texas Medical Center, Houston, Texas
  - Sentara RMH Medical Center, Harrisonburg, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Centro Privado de Cardiología, San Miguel de Tucumán, Argentina
- Australia (6):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital-Clinical Haematology Dept, Westmead, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - St. Vincents Hospital (MEL), Fitzroy, Victoria
- Austria (4):
  - KH der Barmherzigen Schwestern Linz, Linz
  - Kepler Univ. Klinikum Linz, Linz
  - AKH - Medical University of Vienna, Vienna
  - Wilhelminenspital, Vienna
- Belgium (6):
  - Aalst - HOSP Onze-Lieve-Vrouw, Aalst
  - Brussels - UNIV St-Pierre, Brussels
  - Brussels - UNIV UZ Brussel, Brussels
  - Brussels - UNIV St-Luc, Brussels
  - Genk - HOSP ZOL (St-Jan), Genk
  - UZ Leuven, Leuven
- Hospital Nossa Senhora de Pompéia, Caxias do Sul, Brazil
- Canada (4):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Jewish General Hospital, Montreal, Migration Data
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
- Colombia (4):
  - Fundación Valle del Lili, Cali
  - Centro Médico Imbanaco de Cali S.A., Cali
  - Fundación Cardiovascular de Colombia, Floridablanca
  - Hospital Pablo Tobón Uribe, Medellín
- Czechia (6):
  - University Hospital Brno, Brno
  - Hospital,Neurology Dept,Ceske Budejovice, České Budějovice
  - Hospital Hradec Kralove, Hradec Králové
  - Regional Hospital Liberec, Liberec
  - Univ. Hospital Kralovske Vinohrady, Prague
  - University Hospital Motol, Prague
- Aarhus Universitetshospital, Aarhus C, Denmark
- Finland (5):
  - HUS, Kirurginen päivystysosasto P1P, Meilahti, Helsinki, Helsinki
  - Keski-Suomen keskussairaala, Jyväskylä
  - Oulun yliopistollinen keskussairaala, Oulu
  - TAYS, Acuta, Tampere, Tampere
  - TYKS, Akuutti sisätautihoito ASIS, Turku, Turku
- France (11):
  - HOP Trousseau, Chambray-lès-Tours
  - HOP Bocage, Dijon
  - HOP André Mignot, Le Chesnay
  - HOP Lille, SAMU 59, Lille, Lille
  - HOP Dupuytren, Limoges
  - HOP Herriot, Lyon
  - HOP Lapeyronie, Montpellier
  - HOP Haut-Lévêque, Pessac
  - HOP Lyon Sud, Pierre-Bénite
  - HOP Nord, Saint-Priest-en-Jarez
  - HOP Sainte Anne, Urgence, Toulon, Toulon
- Germany (3):
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Hong Kong (3):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Prince of Wales Hosp, Dept of Med & Therapeutics, Hong Kong
- India (2):
  - B.M. Birla Heart research Centre, Kolkata
  - Fortis Escorts Heart Institute, New Delhi
- Ireland (2):
  - St James's Hospital, Dublin
  - Cork University Hospital, Wilton
- Israel (4):
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - The Chaim Sheba Medical Center Tel Hashomer, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Azienda Ospedaliera Careggi, Florence
  - Ospedale S.Maria della Misericordia, AO di Perugia, Perugia
  - Azienda Unità Sanitaria Locale di Reggio Emilia, Reggio Emilia
  - Policlinico Gemelli, Roma
  - Az. Osp. S.Giovanni-Addolorata, Roma
- Japan (12):
  - Japanese Red Cross Nagoya Daini Hospital, Aichi, Nagoya
  - Ehime Prefectural Central Hospital, Ehime, Matsuyama
  - Fukuoka Tokushukai Medical Center, Fukuoka, Kasuga
  - Ogaki Municipal Hospital, Gifu, Ogaki
  - National Hospital Organization Takasaki General Medical Center, Gunma, Takasaki
  - Hyogo College of Medicine Hospital, Hyogo, Nishinomiya
  - National Hospital Organization Kagoshima Medical Center, Kagoshima, Kagoshima
  - Shonan Kamakura General Hospital, Kanagawa, Kamakura
  - National Cerebral and Cardiovascular Center, Osaka, Suita
  - Nippon Medical School Hospital, Tokyo, Bunkyo-Ku
  - National Hospital Organization Disaster Medical Center, Tokyo, Tachikawa
  - Yamagata City Hospital SAISEIKAN, Yamagata, Yamagata
- Hospital Cardiologica Aguascalientes, Aguascalientes, Mexico
- Netherlands (6):
  - OLVG, locatie Oosterpark, Amsterdam
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Martini Ziekenhuis, Groningen
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- New Zealand (5):
  - Christchurch Hospital, Christchurch
  - Auckland City Hospital, Grafton / Auckland
  - Waikato Hospital, Hamilton
  - Middlemore Hospital, Otahuhu South Auckland
  - North Shore Hospital, Takapuna, Takapuna Auckland
- Norway (5):
  - Haukeland Universitetssykehus, Bergen
  - Vestre Viken HF, Drammen Sykehus, Drammen
  - Sykehuset Østfold Kalnes, Grålum
  - Oslo Universitetssykehus HF, Ullevål sykehus, Oslo
  - Universitetssykehuset Nord-Norge, Tromsø, Tromsø
- Poland (8):
  - Univ. Clinic Hosp, Bialystok, Bialystok
  - University Clinical Center, Gdansk, Gdansk
  - Saint Wincenty a Paulo Hosp., Cardiology Dept., Gdynia, Gdynia
  - Reg.Hosp Kielce,Swietokrzyskie,1.Clinic of Cardiology,Kielce, Kielce
  - The John Paul II Hosp.,Dept.of Coronary Heart Disease,Krakow, Krakow
  - Stefan Kardynal Wyszynski Reg.Hosp,Cardiol&IntensUnit,Lublin, Lublin
  - Independent Public Healthcare, Dept. of Cardiology, Pulawy, Puławy
  - Central Hosp.Minis.Interior,Dep.Noninvasive Cardiol,Warszawa, Warsaw
- Portugal (4):
  - Centro Hospitalar da Cova da Beira Hospital Pêro da Covilhã, Covilha
  - CHLO, EPE - Hospital S. Francisco Xavier, Lisbon
  - Centro Hospitalar do Porto, EPE, Porto
  - Centro Hospitalar São João,EPE, Porto
- Russia (2):
  - Military Medical Academy n.a. S. M. Kirov, St. Petersburg, Saint Petersburg
  - City Pokrovskiy Hospital, Cardiology Dept., Saint Petersburg, Saint Petersburg
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore
- South Africa (2):
  - Dr. D. Adler, Sandton
  - Dr. Engelbrecht, Somerset West
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
- Spain (14):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Politècnic La Fe, Valencia
  - Hospital Clínico de Valencia, Valencia
  - Hospital Álvaro Cunqueiro, Vigo (Pontevedra)
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Sweden (3):
  - Sahlgrenska US, Göteborg, Gothenburg
  - Skånes universitetssjukhus, Lund
  - Akademiska sjukhuset, Uppsala
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipe Veterans General Hospital, Taipei
- United Kingdom (7):
  - North Hampshire Hospital, Basingstoke
  - Royal Liverpool University Hospital, Liverpool
  - Royal London Hospital, London
  - St George's Hospital, London
  - Emergency Department, John Radcliffe Hospital, Oxford, Oxford
  - Southampton General Hospital, Southampton
  - Musgrove Park Hospital, Taunton

REFERENCES:
- [Derived] Eikelboom JW, van Ryn J, Reilly P, Hylek EM, Elsaesser A, Glund S, Pollack CV, Weitz JI. Dabigatran Reversal With Idarucizumab in Patients With Renal Impairment. J Am Coll Cardiol. 2019 Oct 8;74(14):1760-1768. doi: 10.1016/j.jacc.2019.07.070. PMID 31582135
- [Derived] Glund S, Coble K, Gansser D, Stangier J, Hoermann K, Pollack CV, Reilly P. Pharmacokinetics of idarucizumab and its target dabigatran in patients requiring urgent reversal of the anticoagulant effect of dabigatran. J Thromb Haemost. 2019 Aug;17(8):1319-1328. doi: 10.1111/jth.14476. Epub 2019 Jun 18. PMID 31050868
- [Derived] Van der Wall SJ, Lopes RD, Aisenberg J, Reilly P, van Ryn J, Glund S, Elsaesser A, Klok FA, Pollack CV Jr, Huisman MV. Idarucizumab for Dabigatran Reversal in the Management of Patients With Gastrointestinal Bleeding. Circulation. 2019 Feb 5;139(6):748-756. doi: 10.1161/CIRCULATIONAHA.118.036710. PMID 30586692
- [Derived] Pollack CV Jr, Reilly PA, van Ryn J, Eikelboom JW, Glund S, Bernstein RA, Dubiel R, Huisman MV, Hylek EM, Kam CW, Kamphuisen PW, Kreuzer J, Levy JH, Royle G, Sellke FW, Stangier J, Steiner T, Verhamme P, Wang B, Young L, Weitz JI. Idarucizumab for Dabigatran Reversal - Full Cohort Analysis. N Engl J Med. 2017 Aug 3;377(5):431-441. doi: 10.1056/NEJMoa1707278. Epub 2017 Jul 11. PMID 28693366
- [Derived] Pollack CV Jr, Reilly PA, Eikelboom J, Glund S, Verhamme P, Bernstein RA, Dubiel R, Huisman MV, Hylek EM, Kamphuisen PW, Kreuzer J, Levy JH, Sellke FW, Stangier J, Steiner T, Wang B, Kam CW, Weitz JI. Idarucizumab for Dabigatran Reversal. N Engl J Med. 2015 Aug 6;373(6):511-20. doi: 10.1056/NEJMoa1502000. Epub 2015 Jun 22. PMID 26095746
- [Derived] Pollack CV Jr, Reilly PA, Bernstein R, Dubiel R, Eikelboom J, Glund S, Huisman MV, Hylek E, Kam CW, Kamphuisen PW, Kreuzer J, Levy JH, Sellke F, Stangier J, Steiner T, Wang B, Weitz JI. Design and rationale for RE-VERSE AD: A phase 3 study of idarucizumab, a specific reversal agent for dabigatran. Thromb Haemost. 2015 Jul;114(1):198-205. doi: 10.1160/TH15-03-0192. Epub 2015 May 28. PMID 26020620

RESULTS

PARTICIPANT FLOW:
Groups:
- Idarucizumab (Group A): Patients who were treated with dabigatran and who had uncontrolled or life threatening bleeding that required urgent medical or surgical intervention were administered idarucizumab 5 g (two 2.5 g vials) as an intravenous (IV) infusion. A single vial contains 2.5 g of idarucizumab. Patients received a 2.5 g vial of study medication and a second 2.5-g vial within the next 15 minutes.
- Idarucizumab (Group B): Patients who were treated with dabigatran and who may not have been bleeding, but required an emergency surgery or other invasive procedure for a condition other than bleeding where therapeutic anticoagulation might have increased the risk of intra- and post-operative bleeding were administered idarucizumab 5 g (two 2.5 g vials) as an intravenous (IV) infusion. A single vial contains 2.5 g of idarucizumab. Patients received a 2.5 g vial of study medication and a second 2.5-g vial within the next 15 minutes.
Period: Overall Study
Arm/Group | Idarucizumab (Group A) | Idarucizumab (Group B)
Started | 301 | 202
Completed | 222 | 146
Not Completed | 79 | 56
Not completed — Withdrawal by Subject | 10 | 3
Not completed — Lost to Follow-up | 4 | 4
Not completed — Protocol Violation | 6 | 8
Not completed — Adverse Event | 57 | 38
Not completed — Other than stated above | 2 | 3

BASELINE CHARACTERISTICS:
Population: Treated set: Treated Set is defined as all patients who were administered idarucizumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Idarucizumab (Group A) | Idarucizumab (Group B) | Total
Number analyzed (Participants) | 301 | 202 | 503
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.1 (10.4) | 75.9 (10.5) | 76.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 100 | 229
  Male | 172 | 102 | 274

OUTCOME MEASURES:

1. Primary Outcome: Maximum Reversal of Anticoagulant Effect of Dabigatran Based on Central Laboratory Determination of dTT or ECT
Description: Maximum reversal of anticoagulant effect of dabigatran based on central laboratory determination of diluted thrombin time (dTT) or ecarin clotting time (ECT), at any time point from the end of the first infusion up to 4 hours after the last infusion.
  Reversal is defined for patients with at least one post-dose coagulation test results and pre-dose result higher than 100% ULN (evaluable patients).
  Reversal is calculated as 100* (pre-dose value minus post dose value)/(pre-dose value minus 100% x ULN); if calculated reversal is > 100, it was set to 100.
Time Frame: from the end of the first infusion up to 4 hours after the last infusion on Day 1
Population: Treated Set
Measure: Median (95% Confidence Interval); unit: percentage
Arm/Group | Idarucizumab (Group A) | Idarucizumab (Group B)
Number analyzed (Participants) | 301 | 202
percentage
  dTT (# patients evaluable for reversal=244; 152) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  ECT (# patients evaluable for reversal=276; 185) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

2. Secondary Outcome: Reversal of aPTT and TT From Central Laboratory
Description: Reversal of anticoagulation as measured by Activated Partial Thromboplastin Time (aPTT) and Thrombin time (TT), at any time point since the end of first infusion up to 4 hours after the completion of the last infusion. Reversal is defined for patients with at least one post-dose coagulation test results and pre-dose result higher than 100% ULN (evaluable patients).
  Reversal is calculated as 100* (pre-dose value minus post dose value)/(pre-dose value minus 100% x ULN); if calculated reversal is > 100, it was set to 100.
Time Frame: from the end of the first infusion up to 4 hours after the last infusion on Day 1
Population: Treated Set
Measure: Median (95% Confidence Interval); unit: percentage
Arm/Group | Idarucizumab (Group A) | Idarucizumab (Group B)
Number analyzed (Participants) | 301 | 202
percentage
  aPTT (# patients evaluable for reversal=232; 141) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  TT (# patients evaluable for reversal=278; 188) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

3. Secondary Outcome: Duration of Reversal
Description: Duration of reversal, defined as the time period a patient remained completely reversed based on dTT or ECT, up to 24 hours or re-starting the treatment of dabigatran.
Time Frame: from the first infusion up to 24 hours after the last infusion on Day 1
Population: Treated Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Idarucizumab (Group A) | Idarucizumab (Group B)
Number analyzed (Participants) | 301 | 202
hours
  ECT (# patients evaluable for reversal=276; 185) | 13.2 (10.0) | 12.8 (9.7)
  dTT (# patients evaluable for reversal=244; 152) | 19.8 (6.7) | 18.8 (7.6)

4. Secondary Outcome: Occurrence of Major/Life-threatening/Fatal Bleeding (for Group B Only) Intraoperatively
Description: Occurrence of major/life-threatening/fatal bleeding (for group B only) intraoperatively and up to 24 hours post-surgery were classified according to major or life-threatening bleeding (ISTH [International Society for Thrombosis and Hemostasis] definition). 95% Confidence Interval (CI) is from Clopper-Pearson method.
Time Frame: within 24 hours of surgery
Population: Treated Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idarucizumab (Group B)
Number analyzed (Participants) | 202
percentage of participants | 3.0 [1.1 to 6.5]

5. Secondary Outcome: Time to Cessation of Bleeding (for Group A Only)
Description: Time to cessation of bleeding (for Group A only) since first infusion up to 24 hours after the completion of second infusion; bleeding status was to be categorized before and at several time points after treatment.
Time Frame: from the first infusion up to 24 hours after the last infusion on Day 1
Population: Treated set with patients who stopped bleeding within 24 hours
Measure: Median (95% Confidence Interval); unit: hours
Groups:
- ICH (Group A): Group A patients with baseline intracranial hemorrhage (ICH).
- Non-ICH (Group A): Group A patients with baseline non-intracranial hemorrhage (non-ICH).
Arm/Group | ICH (Group A) | Non-ICH (Group A)
Number analyzed (Participants) | 41 | 134
hours | 10.73 [4.80 to 15.73] | 2.49 [2.18 to 3.93]

6. Secondary Outcome: Cmin,1 of Unbound Sum (Free) Dabigatran
Description: Cmin,1 (Minimum concentrations at any time point since the end of first vial of idarucizumab up to 4 hours after the completion of second vial) of unbound sum (free) dabigatran, provided that two vials given not more than 15 min apart in group A and B.
Time Frame: Since the end of first vial of idarucizumab up to 4 hours after the completion of second vial
Population: The Pharmacokinetic Set (PKS): This analysis set was used for all PK analyses and was defined as all patients in the Treated Set who provided at least one PK data point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Idarucizumab (Group A & B): In Group A the patients who were treated with dabigatran and who had uncontrolled or life threatening bleeding that required urgent medical or surgical intervention were administered idarucizumab 5 g (two 2.5 g vials) as an intravenous (IV) infusion. A single vial contains 2.5 g of idarucizumab. Patients received a 2.5 g vial of study medication and a second 2.5-g vial within the next 15 minutes.
  In Group B the patients who were treated with dabigatran and who may not have been bleeding, but required an emergency surgery or other invasive procedure for a condition other than bleeding where therapeutic anticoagulation might have increased the risk of intra- and post-operative bleeding were administered idarucizumab 5 g (two 2.5 g vials) as an intravenous (IV) infusion. A single vial contains 2.5 g of idarucizumab. Patients received a 2.5 g vial of study medication and a second 2.5-g vial within the next 15 minutes.
Arm/Group | Idarucizumab (Group A & B)
Number analyzed (Participants) | 493
ng/mL | 1.12 (61.2)

7. Secondary Outcome: Reversal of Anticoagulation as Measured by Diluted Thrombin Time (dTT) or Ecarin Clotting Time (ECT) After the First Vial of Idarucizumab and Before the Start of Second Vial
Description: Reversal of anticoagulation as measured by diluted Thrombin Time (dTT) or Ecarin Clotting Time (ECT) after the first vial of idarucizumab and before the start of second vial.
  Reversal is defined for patients with at least one post-dose coagulation test results and pre-dose result higher than 100% ULN (evaluable patients). Reversal is calculated as 100*(pre-dose value minus post dose value)/(pre-dose value minus 100% x ULN); if calculated reversal is > 100, it was set to 100.
Time Frame: after the first vial of idarucizumab and before the start of second vial on Day1
Population: Treated Set
Measure: Median (95% Confidence Interval); unit: percentage
Arm/Group | Idarucizumab (Group A) | Idarucizumab (Group B)
Number analyzed (Participants) | 301 | 202
percentage
  dTT (# patients evaluable for reversal=240; 150) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  ECT (# patients evaluable for reversal=271; 182) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

ADVERSE EVENTS:
Time Frame: From the first vial of idarucizumab until end of study (90 ± 7 days after the second vial).
Arm/Group | Idarucizumab (Group A) | Idarucizumab (Group B)
Serious Adverse Events (participants affected / at risk) | 160/301 | 106/202
Other Adverse Events (participants affected / at risk) | 139/301 | 86/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idarucizumab (Group A) (N=301) | Idarucizumab (Group B) (N=202)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac amyloidosis (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 9
Cardiac failure (Cardiac disorders) | 11 | 4
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 10 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 2
Coronary artery disease (Cardiac disorders) | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Thyroid haemorrhage (Endocrine disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 2 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 2
Gastrointestinal mucosal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Ileal ulcer (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Adhesion (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 2 | 2
Multiple organ dysfunction syndrome (General disorders) | 2 | 4
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 1 | 0
Medical device site joint infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 14 | 7
Pneumonia bacterial (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 7 | 5
Septic shock (Infections and infestations) | 2 | 11
Urinary tract infection (Infections and infestations) | 6 | 0
Urosepsis (Infections and infestations) | 1 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Stoma site irritation (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 9 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Starvation (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Genital neoplasm malignant female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Brain stem haemorrhage (Nervous system disorders) | 1 | 0
Brain stem syndrome (Nervous system disorders) | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Chorea (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 0 | 1
Intracranial mass (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 5 | 2
Monoplegia (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 1
Simple partial seizures (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Device loosening (Product Issues) | 0 | 1
Delirium (Psychiatric disorders) | 13 | 8
Hallucinations, mixed (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 6
Anuria (Renal and urinary disorders) | 3 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 3
Renal failure (Renal and urinary disorders) | 1 | 5
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 7 | 3
Haematoma (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 2
Shock (Vascular disorders) | 0 | 2
Shock haemorrhagic (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idarucizumab (Group A) (N=301) | Idarucizumab (Group B) (N=202)
Anaemia (Blood and lymphatic system disorders) | 13 | 11
Constipation (Gastrointestinal disorders) | 33 | 20
Diarrhoea (Gastrointestinal disorders) | 14 | 18
Nausea (Gastrointestinal disorders) | 21 | 18
Oedema peripheral (General disorders) | 17 | 14
Pyrexia (General disorders) | 23 | 6
Urinary tract infection (Infections and infestations) | 35 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 8
Dizziness (Nervous system disorders) | 9 | 11
Headache (Nervous system disorders) | 27 | 6
Confusional state (Psychiatric disorders) | 8 | 13
Haematuria (Renal and urinary disorders) | 18 | 6
Hypotension (Vascular disorders) | 17 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.